# **CONSENT FORMS**

# INCREASING PARENT DEMAND FOR EVIDENCE-BASED PRACTICES TO TREAT YOUTH ANXIETY: THE EFFECT OF PARENT KEY OPINION LEADERS

Margaret E. Crane, Marc S. Atkins, Sara J. Becker, Jonathan Purtle, Thomas M. Olino, & Philip C. Kendall

NCT04929262

Secondary ID: 1F31MH124346-01

**February 5, 2021** 



#### **Department of Psychology**

# Temple IRB Approved

02/05/2021

#### CONSENT FORM

**Title of research study:** Project CHAT: Caregivers Hearing about Anxiety Treatments

# **Investigator and Department:**

Principal Investigator: Philip C. Kendall, Ph.D., ABPP

Co-Investigator: Margaret E. Crane, M.A.

Department of Psychology

# Why am I being invited to take part in this research?

We invite you to take part in a research study because you are a parent/caregiver interested in learning more about youth anxiety disorders.

#### What should I know about this research?

- \* Someone will explain this research to you.
- \* Whether or not you take part is up to you.
- \* You can choose not to take part.
- \* You can agree to take part and later change your mind.
- \* Your decision will not be held against you.
- \* You can ask all the questions you want before you decide.

## Who can I talk to about this research?

If you have questions, concerns, or complaints, or think the research has hurt you, contact the research team at pkendall@temple.edu or 215-204-7165.

This research has been reviewed and approved by an Institutional Review Board. You may talk to them at (215) 707-3390 or e-mail them at: irb@temple.edu for any of the following:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

# Why is this research being done?

The purpose of this research is to compare different approaches for providing information about youth anxiety to caregivers. Caregivers have distinct preferences for how they receive information about their child's mental health. This study will see if caregivers find certain approaches more helpful in receiving this information. We will do this by providing caregivers with an educational presentation on youth anxiety. Presentations will take place via Zoom and will be coordinated through your child's school. Participation in this study also will give caregivers the opportunity to ask questions about youth anxiety and seeking effective treatment for anxiety disorders.

## How long will I be in this research?

We expect that you will be involved in this research for approximately three months. The presentation will take 90 minutes. Before and after the presentation, you will complete questionnaires online. Three months after the presentation, all participants will be asked to complete a brief (approximately 15 minutes) questionnaire. We will select 40 participants (20 from each presentation format) to tell us more about your experience in the study during a 30-minute interview 3 months after the presentation. Total expected participation time is approximately 2.75 hours, and 3.25 hours if you participate in the additional interview.

## How many people will be in this research?

We expect about 180 people will take part in this research.

## What happens if I agree to be in this research?

If you agree to participate in this study, you will be asked to attend a virtual 90 minute presentation on youth anxiety. These presentations will take place via Zoom and will be organized through your child's school. There will be two types of presentation, both of which will provide information on identifying anxiety disorders, strategies for caregivers to help their child/teen's with anxiety, effective strategies to treat youth anxiety, and strategies for finding a therapist who uses evidence-based treatments. However, one type of presentation will be presented by two researchers. The other type will be presented by a researcher and a caregivers from your community. The type of presentation you receive was determined in random or chance fashion (like flipping a coin) and is not based on any information you have provided. Neither you nor the research team chose what presentation you receive. You have an equal chance of being in each presentation group.

Immediately before and after the presentation, you will be asked to complete online measures that include questions about your knowledge of effective strategies to treat anxiety, your perception of stigma of mental illness, your opinions about seeking treatments based on research, your child's anxiety symptoms, and your experiences with mental health treatment. You do not have to answer any questions that make you feel uncomfortable. Most caregivers should be able to complete these measures in approximately 60 minutes total. Three months after the presentation, you will be sent a link to complete a brief (8 question) questionnaire. If you are selected to participate in the 30-minute interview, 3 months after the presentation, you will receive an email from the researcher inviting you to complete the interview. In the interview, you will be asked to tell us more about what you thought of the presentation you received, as well as your thoughts about seeking therapy for your child. This interview will take place via Zoom and will be recorded.

## What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible for attending the 90 minute presentation and completing questionnaires when you receive them by e-mail. You also will be responsible for completing the Zoom interview if you are selected.

## What other choices do I have besides taking part in this research?

Instead of being in this research, your choices may include seeking information about youth anxiety online, from another health care provider, or from your school.

## What happens if I agree to be in this research, but I change my mind later?

If you agree to take part in the research now and change your mind, it will not be held against you. However, because the presentation is part of the research, you would no longer be able to attend.

## Is there any way being in this research could be bad for me?

There is minimal risk associated with this research project. Some caregivers may feel distressed should they realize that their child has an anxiety disorders, or from completing questionnaires about their experience with mental health treatment. However, the presentation aims to increase the caregiver's ability to seek psychological treatment for their youth, so the risk of presentation-related distress is minimal. There is a risk of loss of confidentiality. Time burden is another potential risk.

## Will being in this research help me in any way?

As part of this study, you will receive information about child anxiety and how to seek treatment for child anxiety at no cost.

## What happens to the information we collect for this research?

To the extent allowed by law, we limit the viewing of your personal information to people who have to review it. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB, Temple University, the National Institute of Mental Health, and the Office of Human Research Protections.

Even though the study team has put safeguards in place to protect your information, there is always a potential risk of loss of confidentiality. The identifying information that will be seen by the research team and may be collected includes your name, address, and email address. To help ensure confidentiality, information that is collected for this research will be identified by a unique ID. REDCap (the survey collection software we use) is HIPAA compliant. We will also make sure to store information collected for the research so that only the research team will be able to access it.

We may publish the results of this research. However, we will keep your name and other identifying information entirely confidential. Information is reported without naming anyone in the study.

## What if I am injured because of taking part in this research?

If you are injured as a result of taking part in this research, immediately notify the research team and they will arrange for you to get immediate medical care. There is no commitment by Temple University, Temple University Health System or its subsidiaries to provide monetary compensation or free medical care to you in the event of a research-related injury. If you have a research-related injury, please contact Dr. Kendall at (215) 204-7165 during regular hours and at (215) 694-5546 after hours and on weekends and holidays.

# What will I be paid for taking part in this research?

If you agree to take part in this research, we will pay you \$20 for attending the presentation and completing questionnaires before and after the presentation. You must complete the post-presentation questionnaires within 1 week of the presentation to receive payment. You will be paid \$10 for completing the 3 month follow-up survey. If you are asked to complete another 30-minute interview at the end of the study, you will receive an additional \$20. All payments will be in the form of a visa gift card.

Federal tax law requires to you to report this payment as income to the Internal Revenue Service. You may be asked to tell us your social security number, full name, address, or other identifying information in order to compensate you for your participation. We may request this is because we are required to report payments more than \$599.00, to the Internal Revenue Service and you will be sent a Form 1099-MISC.

| Your signature documents your permission to take part in this research. | |
|---|---|
| Signature of subject | Date |
| Printed name of subject | <u>—</u> |



#### **Department of Psychology**

Temple IRB Approved

02/05/2021

#### CONSENT FORM

**Title of research study:** Project CHAT: Caregivers Hearing about Anxiety Treatments

## **Investigator and Department:**

Principal Investigator: Philip C. Kendall, Ph.D., ABPP

Co-Investigator: Margaret E. Crane, M.A.

Department of Psychology

# Why am I being invited to take part in this research?

We invite you to take part in a research study because you are a parent who has been identified as a key opinion leader by your parent teacher association.

#### What should I know about this research?

- \* Someone will explain this research to you.
- \* Whether or not you take part is up to you.
- \* You can choose not to take part.
- \* You can agree to take part and later change your mind.
- \* Your decision will not be held against you.
- \* You can ask all the questions you want before you decide.

#### Who can I talk to about this research?

If you have questions, concerns, or complaints, or think the research has hurt you, contact the research team at pkendall@temple.edu or 215-204-7165.

This research has been reviewed and approved by an Institutional Review Board. You may talk to them at (215) 707-3390 or e-mail them at: irb@temple.edu for any of the following:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

# Why is this research being done?

The purpose of this research is to compare different approaches for providing information about youth anxiety to caregivers. Caregivers have distinct preferences for how they receive information about their child's mental health. This study will see if caregivers find certain approaches more helpful in receiving this information. We will do this by providing caregivers with an educational presentation on youth

anxiety. Participation in this study also will give caregivers the opportunity to ask questions about youth anxiety and seeking effective treatment for anxiety disorders.

# How long will I be in this research?

We expect that you will be involved in this research for at least 1 month. Your involvement will include a two-hour focus group, a 1 hour Zoom call with the researcher, and attending the two-hour presentation. You also may wish to spend additional time preparing for the presentation. The focus groups will occur at least 1 month prior to the presentation at the schools. The exact timing will depend on the school's schedule.

## How many people will be in this research?

We expect about 4 other caregivers to participate as a co-presenter in this research.

## What happens if I agree to be in this research?

If you agree to participate in this study, you will be asked to attend a two-hour training with at least one other caregiver co-presenters. Before the training, you will be asked to complete a questionnaire about your demographic information. You do not have to answer any questions that make you feel uncomfortable. You also will be sent the presentation to review before the training.

During the training, you will discuss your experiences with youth anxiety, factors about your communities that may affect how anxiety symptoms present or are understood, and how caregivers in your community typically seek therapy. You also will be asked to consider which strategies you can endorse as being effective (e.g., remaining calm when their child becomes emotional). We will review the presentation materials and encourage you to discuss your reactions and provide feedback. Following the training, we will meet with each you presenter individually via phone to (1) review/approve the modifications made; (2) answer remaining questions about the content; (3) determine which sections you are comfortable presenting, and which strategies you are willing to endorse; and (4) give you an opportunity to practice to ensure comprehension. Finally, you will present a portion of the 90 minute presentation for caregivers at your school. Please allot 2 hours to attend the outreach presentation.

## What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible for attending the two-hour training, the follow-up phone call, co-presenting information to caregivers, and completing the demographic questionnaire.

## What other choices do I have besides taking part in this research?

Instead of being in this research, your choices include attending attend the educational presentation at your school as a participant; seeking information about youth anxiety online, from another health care provider, or from your school; or not participating in any other form.

## What happens if I agree to be in this research, but I change my mind later?

If you agree to take part in the research now and change your mind, it will not be held against you.

## Is there any way being in this research could be bad for me?

There is minimal risk associated with this research project. Some caregivers may feel distressed should they realize that their child has an anxiety disorders, or from completing questionnaires about their experience with mental health treatment. However, the presentation aims to increase the caregiver's ability to seek psychological treatment for their youth, so the risk of presentation-related distress is minimal. There is a risk of loss of confidentiality. Time burden is another potential risk.

## Will being in this research help me in any way?

As part of this study, you will receive information about child anxiety and how to seek treatment for child anxiety at no cost.

# What happens to the information we collect for this research?

To the extent allowed by law, we limit the viewing of your personal information to people who have to review it. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB, Temple University, the National Institute of Mental Health, and the Office of Human Research Protections.

Even though the study team has put safeguards in place to protect your information, there is always a potential risk of loss of confidentiality. The identifying information that will be seen by the research team and may be collected includes your name, address, and email address. To help ensure confidentiality, information that is collected for this research will be identified by a unique ID. REDCap (the survey collection software we use) is HIPAA compliant. We will also make sure to store information collected for the research so that only the research team will be able to access it.

We may publish the results of this research. However, we will keep your name and other identifying information entirely confidential. Information is reported without naming anyone in the study.

## What if I am injured because of taking part in this research?

If you are injured as a result of taking part in this research, immediately notify the research team and they will arrange for you to get immediate medical care. There is no commitment by Temple University, Temple University Health System or its subsidiaries to provide monetary compensation or free medical care to you in the event of a research-related injury. If you have a research-related injury, please contact Dr. Kendall at (215) 204-7165 during regular hours and at (215) 694-5546 after hours and on weekends and holidays.

# What will I be paid for taking part in this research?

If you agree to take part in this research, we will pay you \$200 (in the form of a visa gift card) after the presentation for your time and efforts.

Federal tax law requires to you to report this payment as income to the Internal Revenue Service. You may be asked to tell us your social security number, full name, address, or other identifying information in order to compensate you for your participation. We may request this is because we are required to report payments more than \$599.00, to the Internal Revenue Service and you will be sent a Form 1099-MISC.

| Your signature documents your permission to take part in this research. | |
|---|---|
| Signature of subject | Date |
| Printed name of subject | |